CLINICAL TRIAL: NCT00981344
Title: Wheeled Mobility in Everyday Life: Effects of Wheelchair Type on Mobility Performance of Elders in Public Environments
Brief Title: Wheeled Mobility in Everyday Life
Acronym: RERC-4a
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Pro00012299; NIDRR, H133E80003
Record Dates: First submitted 2009-09-15; First posted 2009-09-22 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Heart Disorder; Lung Disorder; Arthritis
Keywords: wheelchair; mobility disability; evidence based practice; self help devices; Veterans prescribed mobility aids
MeSH Terms: conditions — Lung Diseases; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Wheeled Mobility in Everyday Life:Effects of Wheelchair Type on Mobility Performance of Elders in Public Environments — We are studying how wheeled mobility performance and the impact of device type on a group of community dwelling Veterans.
  Other Names: RERC-4a; Wheeled Mobility in Everyday Life

SUMMARY:
The project will examine how mobility performance in real life tasks and environments is impacted by the use of specific types of wheeled mobility devices (wheeled walker, manual wheelchair, power wheelchair/scooter). Specifically, the project will: 1) randomly recruit persons who were prescribed a mobility aid within the preceding 1 year and currently use the mobility aid, 2) define key mobility tasks within a public environment, 3) measure mobility performance of subjects as they perform the mobility tasks in each of the four devices, and 4) synthesize and disseminate the results. Study results will be used to establish baseline performance data for researchers and clinicians and to identify design improvements for wheelchairs used by community dwelling elders.

All study participants will be required to complete study related questionnaires about their family environment and familiarity with the various types of mobility aids. In addition, physical abilities will be measured at the start of the study, including measures of arm and leg strength, and the ability to walk and push a wheelchair. This will take about 30 minutes. A total of 150 subjects will be recruited among Veterans prescribed mobility aids in the preceding 3-12 months identified through administrative data sources.

The mobility aids being studied are all standard types of mobility aids used by people with limited mobility (e.g., wheeled walker, manual wheelchair, power wheelchair/scooter). Analyses will proceed in a stepwise fashion. The first step will be to examine the primary study question relating device type to the dependent variable, with velocity being the primary outcome. The next step in the analysis will be to determine if there is an interaction between medical condition, mobility devices, and the dependent variable. Finally, exploratory analyses will be carried out to examine the relationship between baseline measures of physical function and mobility performance with each of the devices. Study related risks are minimal.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed wheeled walker, manual wheelchair, power mobility device in last 3-12 months
* Have chronic heart (e.g., congestive heart failure) or lung disorder (e.g., chronic obstructive pulmonary disease), and/or arthritic disorder (e.g., osteoarthritis)
* Reports using wheeled walker, manual wheelchair, or power mobility device in the preceding 2 weeks

Exclusion Criteria:

* Reports missing one or more limbs and/or complete paralysis of one or more limbs
* Have a neurological, myopathic, or cognitive disorder
* Weight more than 300 lbs; height more than 74 inches
* Poorly controlled hypertension, unstable angina, a heart attack or heart surgery within the last 6 months.
* Reports any of the following: Does not have an active Drivers License, unable to walk across small room without human help, unable to propel w/ch across small room without human help (applies only to those already using a manual w/ch), needs moderate assistance from another person to transfer, unable to sit on side of bed independently, currently has shoulder pain with self care or with wheelchair use.
* Major surgery affecting abdominal, chest, spine, upper extremity in the last 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Speed (in meters/second) | trial duration (generally 1 to 20 minutes)

SECONDARY OUTCOMES:
Self Report of exertion, pain, fatigue,and device preference | completion of study (generally 20 to 40 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Hoenig, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Durham VA Hospital, Durham, North Carolina